CLINICAL TRIAL: NCT03581513
Title: Deferred Versus Immediate Stent Implantation for Preventing Microvascular Dysfunction and Improving Clinical Outcomes in Patients With ST-Segment Elevation Myocardial Infarction (SALVAGE)
Brief Title: Deferred or Immediate Stent Implantation Based on Microvascular Function in STEMI
Acronym: SALVAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB halted the study due to safety concerns.
Sponsor: Harbin Medical University (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Jiamusi City Central Hospital (Unknown); Mudanjiang cardiovascular hospital (Unknown); Shuangyashan Mining Hospital (Unknown); First Affiliated Hospital of Jiamusi University (Unknown); Daqing Longnan Hospital (Unknown); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yu Bo, Clinical Professor, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1301104
Record Dates: First submitted 2018-06-15; First posted 2018-07-10 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Microcirculatory Perfusion; ST Elevation Myocardial Infarction
Keywords: deferred stent implantation; immediate stent implantation; microcirculation function; ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IMR<40 and defer PCI (Experimental): Patients whose IMR<40 undergo stent implantation after an interval of 7±2 days.
  Interventions: Procedure: Deferred or Immediate Stent Implantation
- IMR<40 and immediately PCI (Active Comparator): Patients whose IMR<40 undergo immediately stent implantation.
  Interventions: Procedure: Deferred or Immediate Stent Implantation
- IMR≥40 and defer PCI (Experimental): Patients whose IMR≥40 undergo stent implantation after an interval of 7±2 days.
  Interventions: Procedure: Deferred or Immediate Stent Implantation
- IMR≥40 and immediately PCI (Active Comparator): Patients whose IMR≥40 undergo immediately stent implantation.
  Interventions: Procedure: Deferred or Immediate Stent Implantation

INTERVENTIONS:
Procedure: Deferred or Immediate Stent Implantation — IMR can be used to measure the microcirculatory resistance of coronary artery. It is not clear whether the IMR value could determine the time of PCI for STEMI patients.

SUMMARY:
Timely percutaneous coronary intervention (PCI) with stenting implantation is the current standard treatment for patients with ST-segment elevation myocardial infarction (STEMI). However, stenting in thrombus-laden artery is associated with higher risk of embolization and no-or slow-reflow, leading to larger infarct size and poor prognosis. The SALVAGE study is a prospective, multicenter, randomized, controlled study aimed to optimize the therapeutic strategies (deferred vs. immediate stenting) to protect microvascular function and eventually improve clinical outcomes at 12-months in STEMI.

DETAILED DESCRIPTION:
Methodology:

A multicenter, prospective, randomized, controlled clinical study enroll patients with ST-segment elevation myocardial infarction (STEMI) intended for PCI with stenting implantation. Eligible patients are randomly assigned to the immediate stenting group or delayed stenting group in a 1:1 ratio when residual stenosis >70% and TIMI grade 3 with angiography guidance.

The index of microcirculation resistance (IMR) is quantitative analysis by an invasive approach for evaluating post-infarct myocardial microcirculatory perfusion. IMR correlates with the infarct size of patients with acute myocardial infarction and predicts the improvement in left ventricular ejection fraction. Studies have shown that acute myocardial infarction patients with IMR >40 after primary PCI predict adverse long-term clinical outcomes with higher mortality and heart failure rehospitalization rates.

According to therapeutic strategies and microvascular function detected by IMR, participants are classified into four groups: immediate stenting with IMR ≥ 40, immediate stenting with IMR < 40, deferred stenting with IMR ≥ 40 and deferred stenting with IMR < 40. All randomized patients will be followed by phone call or clinical visit at 12 months.

Patient enrollment and procedure overview:

Patients aged from 18 to 80 with STEMI<12h in whom PCI is planned will be screened. Thrombectomy and balloon dilatation will be performed at the operator's discretion to restore an effective antegrade blood flow with TIMI flow grade 3. Patients with residual diameter stenosis >70% visually and TIMI blood flow grade 3 are eligible for including in the study. All patients must provide written informed consent and patients will be randomized to immediate stenting group or deferred stenting group in a 1:1 ratio. All participants in immediate stenting group will be treated with stent implantation immediately. Those assigned to the deferred arm will undergo stenting after an interval of 7±2 days. This interval will be bridged with anti-coagulant and anti-platelet therapy to reduce thrombus burden. All patients in both groups are required to take dual antiplatelet treatment while the application of low molecular weight heparin and glycoprotein IIb/IIIa inhibitor are determined by the operators. All participants are required to perform IMR pre-stenting and post-stenting to evaluate microcirculation function. All randomized patients will be followed up to 12 months to evaluate the prevalence of heart failure, all-cause mortality, recurrent infarction or targeted vessel revascularization.

Study follow-up:

Clinical follow-up:

Participants will be followed by phone calls or clinical visits by study coordinators at 1 month (+/-7 days), 3 months (+/-15 days), 6 months (+/-15 days), 9 months (+/-15 days) and 12 months (+/-30 days) after randomization. Major adverse cardiovascular events (MACEs) will be recorded throughout the study period until last patient has been followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 80 years old;
* STEMI and the onset time <12h;
* The culprit lesions are de novo lesion;
* Sign written informed consent.

Exclusion Criteria:

* Patients are hemodynamically unstable;
* Infract-related artery diameter stenosis ≤ 70%;
* Left main disease;
* AMI caused by surgery, trauma, gastrointestinal bleeding or PCI and complications;
* AMI occurs in patients who have been hospitalized for other reasons;
* The investigator judges that the patient has poor compliance and cannot complete the study as required;
* Life expectancy ≤ 12 months;
* Heart transplant patients;
* Definite diagnosis of patients with tumors;
* Participate in other clinical studies (excluding other trials of this project) and haven't reach the primary endpoints.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of heart failure, all-cause death, reinfarction and targeted vessel revascularization within 1 year of STEMI | 1 year
  MACE including the prevalence of heart failure, all-cause death, reinfarction and targeted vessel revascularization will be collected as the primary outcome.

SECONDARY OUTCOMES:
Peri-procedural myocardial reperfusion reinjury | through hospitalization, an average of 7 days
  Prevalence of in-hospital heart failure, all-cause death, re-myocardial infarction or targeted vessel revascularization.
Procedural success and clinical success | postprocedure and through hospitalization, an average of 7 days
  Culprit lesion stenosis<30% in the presence of TIMI 3 grade flow after PCI are regarded as procedural success.
  Clinical success is determined as procedural success in the absence of in-hospital cardiac death, target vessel myocardial infarction and clinically-driven target lesion revascularization.
ECG ST-segment resolution at 90 minutes after primary PCI | 90 minutes postprocedure
  We will compare the differences of the ST-segment resolution at 90 minutes among groups after primary PCI.
Peaks of CK, CK-MB, cTnI and area under CK curve | through hospitalization, an average of 7 days
  We will compare the peaks of CK, CK-MB, cTnI and area under CK curve while in hospital.
LVEF detected by echocardiographic indices at 7 days after stenting, 1 month and 12 months after discharge | 7 days, 1 month and 12months
  LVEF will be detected by echocardiographic indices at 7 days after stenting, 1 month and 12 months after discharge
Contrast score index and myocardial blood flow detected by myocardial contrast echocardiography 7 days after stenting and 1 month after discharge | 7 days and 1 month
  Contrast score index and myocardial blood flow detected by myocardial contrast echocardiography 7 days after stenting and 1 month after discharge
Hospitalization due to heart failure | 1 year
  Prevalence of hospitalization for heart failure will be compared among groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, Study Chair — The Second Affiliated Hospital of Harbin Medical University; Xinshun Gu, Principal Investigator — The Second Hospital of Hebei Medical University; Lixin Lu, Principal Investigator — Daqing Longnan Hospital; Zhiyuan Weng, Principal Investigator — Jiamusi City Central Hospital; Kai Liu, Principal Investigator — Mudanjiang cardiovascular hospital; Hui Li, Principal Investigator — Shuangyashan Mining Hospital; Shan Gao, Principal Investigator — First Affiliated Hospital of Jiamusi University; ChunMei Wang, Principal Investigator — Beijing An Zhen Hospital, Capital Medical University
Locations (8):
- China (8):
  - Beijing An Zhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Second hospital of hebei medical university, Shijiazhuang, Hebei
  - Daqing Longnan Hospital, Daqing, Heilongjiang
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiamusi City Central Hospital, Jiamusi, Heilongjiang
  - The First Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - Mudanjiang Cardiovascular Hospital, Mudanjiang, Heilongjiang
  - Shuangyashan Mining Hospital, Shuangyashan, Heilongjiang

REFERENCES:
- [Derived] Feng X, Xu Y, Zeng M, Qin Y, Weng Z, Sun Y, Gao Z, He L, Zhao C, Wang N, Zhang D, Wang C, Wang Y, Li L, Fang C, Dai J, Jia H, Yu B. Optical Coherence Tomography Assessment of Coronary Lesions Associated With Microvascular Dysfunction in ST-Segment Elevation Myocardial Infarction. Circ J. 2023 Oct 25;87(11):1625-1632. doi: 10.1253/circj.CJ-23-0200. Epub 2023 Sep 6. PMID 37407487